CLINICAL TRIAL: NCT06638892
Title: Cluster Randomized Controlled Trial of Using PrEP, Doing it for Ourselves [UPDOs] Protective Styles: A Multi-level Intervention to Improve HIV Testing and PrEP Uptake Among At-risk Populations Living in the Southeastern Region of the United States
Brief Title: Using PrEP, Doing It for Ourselves
Acronym: UPDOs
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00116215; 1R01NR021692 (NIH)
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-02

CONDITIONS: HIV Prevention; PrEP
Keywords: Black Women; Community-based Research
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Using PrEP, Doing it for Ourselves (UPDOs) intervention (Experimental): This group will receive the UPDOs intervention that includes "edutainment", e.g., videos, blogs, vlogs, and Q Care Plus.
  Interventions: Behavioral: Using PrEP, Doing it for Ourselves (UPDOs)
- Standard of Care (Other): This group will receive CDC standard of care, e.g., CDC videos and website.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Behavioral: Using PrEP, Doing it for Ourselves (UPDOs) — An e-Health intervention that considers women's lived experiences and uses three components: beauty salons and stylists as opinion leaders (trusted gatekeepers who share health information in the community), theory driven edutainment videos and blogs, and a secure online platform for accessing pre-exposure prophylaxis (PrEP).
  Arms: Using PrEP, Doing it for Ourselves (UPDOs) intervention
Other: Standard of Care — CDC standard of care, e.g., CDC videos and website.
  Arms: Standard of Care

SUMMARY:
The goal of this clinical trial is to test a new online program called UPDOs Protective Styles to help people in the southeastern United States learn about and start using PrEP (pre-exposure prophylaxis), a medicine that helps prevent HIV. The study focuses on people who may be at higher risk for HIV and have not had equal access to PrEP.

The main questions it aims to answer are:

Does UPDOs help more people trust and understand PrEP? Does UPDOs increase the number of people who start and continue using PrEP?

Researchers will compare two groups:

One group will use UPDOs, which includes six weekly videos, blog discussions, and access to telehealth services through Q Care Plus. The other group will receive standard HIV prevention materials from the CDC.

Participants will:

Be recruited from 32 beauty salons in areas with high HIV rates. Complete surveys at the start of the study and again at 6, 12, 24, 32, and 52 weeks.

Have access to HIV testing and PrEP prescriptions through Q Care Plus.

This study will also look at how well the program works in different communities and how easy it is to use and share.

DETAILED DESCRIPTION:
HIV disproportionately affects people living in the United States Southeast, threatening progress toward the Ending the HIV Epidemic (EHE) initiative's 2030 goals. Therefore, interventions that consider the lived experiences and needs of this at-risk population are urgently needed to support individuals in these geographic areas from medication precontemplation to uptake to maintenance.

Under the leadership of the Principal Investigator and in partnership with communities, an established Community Advisory Council (CAC), an online telehealth platform (Q Care Plus), and beauty salon stylists, the research team co-developed Using PrEP, Doing it for Ourselves (UPDOs) Protective Styles, an e-Health intervention that strongly considers the unique needs of at-risk individuals. This intervention consists of training for stylists to become opinion leaders (trusted gatekeepers who share health information in the community) in HIV prevention (i.e., PrEP), and a 6-week web-based edutainment video series (six 20-minute episodes), structured debrief blogs, and telehealth service access. The CAC was invaluable in this development process, having collaborated with the research team across sexual health-based projects that informed and contributed to UPDOs preliminary research.

UPDOs web content shares core concepts by telling the stories of at-risk individuals in the US Southeast from various backgrounds and role-plays the PrEP decision-making process. Pilot research conducted by the research team found UPDOs acceptable, improved PrEP trust, increased knowledge-for both PrEP-aware and PrEP-unaware participants-and decreased perceptions of PrEP stigma within personal relationships. This proposed effectiveness-implementation type-I hybrid study will test UPDOs effectiveness in a larger, more geographically diverse sample using a cluster-randomized control trial and examine implementation determinants of UPDOs. In collaboration with Q Care Plus, a secure online platform to access telehealth services for home-delivered HIV testing and PrEP prescriptions, the research team will track how many at-risk individuals within counties of increased HIV infections reach out to a provider, get HIV testing, start PrEP, and maintain PrEP as prescribed.

A cohort of 32 beauty salons will be randomized to either an intervention group (n=16) or control group (n=16). Salons (1 salon = 1 cluster) will be randomized to UPDOs (edutainment videos + blogs + Q Care Plus) or usual care (CDC videos + website) conditions. Once salons are randomized, the recruitment and enrollment period of customers will occur over 24 months. Study participation will include data collection at baseline with follow-up measures at 6, 12, 24, 32, and 52 weeks. To assess implementation outcomes and context, the UPDOs Protective Styles research team will perform a mixed methods approach guided by the Consolidated Framework for Implementation Research (CFIR).

Although pre-exposure prophylaxis [PrEP] (an oral or injectable medication that is effective in preventing HIV) has been effective in decreasing HIV acquisition, PrEP uptake for increasingly at-risk populations in the US Southeast remains low. PrEP uptake is as low as 2% for some at-risk communities due to factors influencing decision-making to take PrEP, such as lack of awareness, distrust, stigma, and access. There is an urgent need to provide specific strategies to improve PrEP uptake in ways that are acceptable and feasible for individuals in the US Southeast. Engaging non-traditional settings, such as beauty salons, is one promising strategy. Additionally, engaging communities of interest is effective in reducing HIV for difficult-to-reach at-risk populations and should be prioritized.

In component two, over 6 weeks, customers will view six edutainment videos that use stories, humor, and drama to highlight relevant messages that include HIV/PrEP. Debrief video blogs will follow each episode to highlight key points. Educational media designed to entertain have been effective in improving HIV prevention messaging.

The long-term goal of the Principal Investigator is to implement a real-world, sustainable intervention that will improve PrEP uptake and be scalable across the US South, where HIV inequalities are pronounced (51%) compared to other regions. For example, new diagnosis rates in North Carolina counties-Cumberland, Durham, Forsyth, Guilford, Mecklenburg, and Wake-where this study will take place, were higher than the state average. Thus, the aims of this study are:

• Aim 1:To test the effectiveness of the UPDOs intervention to improve PrEP uptake for at-risk individuals in the US Southeast using the Motivational PrEP Cascade framework within a community-engaged cluster-randomized controlled trial of intervention (UPDOs; N=16) and control (CDC information; N=16) salon clusters.

Hypothesis: Compared to control salons, salon customers in UPDOs (stylist opinion leaders, edutainment videos + blogs, and Q Care Plus) will have higher PrEP uptake.

* Aim 2: To examine the barriers and facilitators underlying PrEP decision-making among a subsample in both intervention (n=20) and control groups (n=20) using quantitative surveys and qualitative individual interviews.
* Aim 3: To understand the facilitators influencing implementation of UPDOs for future scalability using quantitative surveys and qualitative interviews grounded in the CFIR framework.

This proposed study has the potential to significantly advance EHE goals through an efficacious and cost-effective intervention for individuals in the US Southeast that can be scaled quickly throughout the US South.

The Principal Investigator proposes an effectiveness-implementation type-I hybrid study to test the intervention Using PrEP, Doing it for Ourselves (UPDOs) Protective Styles and its effectiveness to improve PrEP uptake among at-risk communities in the US Southeast using a cluster-randomized control trial and examining implementation determinants of UPDOs for scalability across the US South. Project activities will be delivered by an interdisciplinary research team advised by an external advisory panel and established community advisory council and implemented across six North Carolina counties with high concentrations of HIV incidences: Cumberland, Durham, Forsyth, Guilford, Mecklenburg, and Wake. At the conclusion of the funded project, the Principal Investigator and research team will have rigorously evaluated the intervention, ready for scale-up across the US South, with potential to significantly advance EHE goals for at-risk populations unreached by past HIV prevention efforts.

ELIGIBILITY:
Inclusion Criteria:

* Black
* cisgender female
* Ages 18+

Exclusion Criteria:

* Under 18 years of age
* Does not identify as Black
* Not a cisgender female

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Cisgender females
Enrollment: 1000 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Pre-exposure prophylaxis (PrEP) Contemplation Ladder total score | 12 weeks post-intervention
  The PrEP Contemplation Ladder is a 1-item survey designed to measure Motivational PrEP Cascade (MPC) stages of behavior change that represent one's PrEP intentions by a score of 1-10. Scores correspond to MPC stages. Lower numbers indicate PrEP is not being used to prevent HIV and the participant is not really thinking of ever starting to use PrEP. Higher numbers indicate that PrEP is being used daily and the participant is returning for provider checkups and HIV/STI testing every 3 months, as recommended.

SECONDARY OUTCOMES:
Change in pre-exposure prophylaxis (PrEP) Contemplation Ladder total score - 12 to 24 weeks | 12 to 24 weeks post-intervention
  The PrEP Contemplation Ladder is a 1-item survey designed to measure Motivational PrEP Cascade (MPC) stages of behavior change that represent one's PrEP intentions by a score of 1-10. Scores correspond to MPC stages. Lower numbers indicate PrEP is not being used to prevent HIV and the participant is not really thinking of ever starting to use PrEP. Higher numbers indicate that PrEP is being used daily and the participant is returning for provider checkups and HIV/STI testing every 3 months, as recommended.
Change in pre-exposure prophylaxis (PrEP) Contemplation Ladder total score - 24 to 32 weeks | 24 to 32 weeks post-intervention
  The PrEP Contemplation Ladder is a 1-item survey designed to measure Motivational PrEP Cascade (MPC) stages of behavior change that represent one's PrEP intentions by a score of 1-10. Scores correspond to MPC stages. Lower numbers indicate PrEP is not being used to prevent HIV and the participant is not really thinking of ever starting to use PrEP. Higher numbers indicate that PrEP is being used daily and the participant is returning for provider checkups and HIV/STI testing every 3 months, as recommended.
Change in pre-exposure prophylaxis (PrEP) Contemplation Ladder total score - 32 to 52 weeks | 32 to 52 weeks post-intervention
  The PrEP Contemplation Ladder is a 1-item survey designed to measure Motivational PrEP Cascade (MPC) stages of behavior change that represent one's PrEP intentions by a score of 1-10. Scores correspond to MPC stages. Lower numbers indicate PrEP is not being used to prevent HIV and the participant is not really thinking of ever starting to use PrEP. Higher numbers indicate that PrEP is being used daily and the participant is returning for provider checkups and HIV/STI testing every 3 months, as recommended.

CONTACTS AND LOCATIONS:
Overall Officials: Schenita Randolph, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University School of Nursing, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Only statistical information for primary and secondary outcomes will be shared. Individual participant data will not be shared.

DOCUMENTS (1):
  • Informed Consent Form (2024-11-22): https://cdn.clinicaltrials.gov/large-docs/92/NCT06638892/ICF_001.pdf